CLINICAL TRIAL: NCT02089750
Title: Orthotic Use for Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Orthotic Use for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Health Sciences (Other)
Collaborators: University of Illinois at Chicago (Other); Foot Levelers, Inc. (Industry)
Responsible Party: Principal Investigator, Jerrilyn Cambron, DC, PhD, Professor in the Department of Research, National University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUHS IRB_H-1203
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Chronic Low Back Pain
Keywords: Low Back Pain; Chiropractic; Shoe Orthotics
MeSH Terms: conditions — Low Back Pain | interventions — Braces; Waiting Lists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Orthotics (Active Comparator): Subjects are asked to wear custom-made shoe orthotics for a 12 week study period.
  Interventions: Other: Orthotics
- Orthotics Plus Chiropractic Care (Active Comparator): Subjects are asked to wear custom-made shoe orthotics for a 12 week study period in addition to receiving Chiropractic Care 1-4 times per week during the first 6 weeks of the 12 week study period.
  Interventions: Other: Orthotics; Other: Orthotics Plus Chiropractic Care
- Wait List (Other): The group serves as a cross-over control group. Subjects are asked to avoid any new therapies for the first 6 weeks of the 12 week study and during the last six weeks they are fitted for the custom-made shoe orthotics.
  Interventions: Other: Orthotics; Other: Wait List

INTERVENTIONS:
Other: Orthotics
Other: Orthotics Plus Chiropractic Care — The six week Chiropractic Care portion of this intervention may include the use of ice packs, hot packs, massage, and chiropractic manipulations to the spine or lower extremities (utilizing High Velocity Low Amplitude and/or Flexion Distraction manipulations).
  Arms: Orthotics Plus Chiropractic Care
Other: Wait List
  Arms: Wait List

SUMMARY:
The goal of this randomized clinical study is to assess pain and dysfunction in 225 volunteer subjects who have chronic low back pain.

The hypothesis of this study is that custom-made shoe will improve patients' low back pain and dysfunction. Additionally, custom-made shoe orthotics plus chiropractic treatment will further improve patients' low back pain and dysfunction while maintaining that improvement during the one year study follow-up period.

Specific Aims:

1. To determine the changes in perceived pain levels (Numeric Pain Rating Scale) and dysfunction (Oswestry Disability Index) in patients with chronic low back pain after six weeks of custom-made shoe orthotic use with or without chiropractic care as compared to no care.
2. To determine the changes in perceived pain levels and dysfunction in patients with chronic low back pain after twelve weeks of custom-made shoe orthotic use.
3. To determine the changes in perceived pain levels and dysfunction at 3, 6, and 12 months following the 12 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Subjects must be symptomatic with current pain between T12 and the SI joints with or without radiating pain at an average score of 4 or higher on the NPRS scale
3. Symptoms must have been present for at least three months

Exclusion Criteria:

1. Use of custom-made orthotics in the past 6 months
2. Ongoing active conservative care (such as physical therapy or chiropractic care) for the low back, leg, or foot received in the past 6 months (excluding the use of oral medications or daily at-home exercises for general well-being).
3. Current or future litigation for any healthcare concern
4. Not fluent or literate in the English language. We will not be able to provide multiple translators within this study
5. Brain disorders (e.g., dementia, Alzheimers Disease , etc.) that would lead to difficulty in questionnaire completion
6. Chronic pain other than low back pain, such as fibromyalgia or multiple sclerosis
7. Clinically significant chronic inflammatory spinal arthritis
8. Spinal pathology or fracture
9. Progressive neurologic deficits due to nerve root or spinal cord compression, including symptoms/signs of cauda equina syndrome
10. History of bleeding disorder
11. Known arterial aneurysm
12. Previous lumbar spine surgery
13. Severe skeletal deformity of the foot
14. Peripheral neuropathy due to disorders such as diabetes
15. Low back pain that is not reproducible
16. Current pregnancy
17. Other conditions that may affect the subjects' ability to participate throughout the duration of the study or exclude patients from participation in the study, including contraindications to orthotic use or chiropractic spinal manipulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | This primary outcome measure will be collected at the Randomization Visit and Week 6.
  The Numeric Pain Rating Scale (NPRS) is a numeric scale from 0-10, wherein patients can select (by circling or otherwise selecting) the one number along that line that best describes the pain being inquired about during the specified time period. The NPRS is one of the most frequently used methods for the measurement of clinical pain.
Modified Oswestry Disability Index (MODI) | This primary outcome measure will be collected at the Randomization Visit and Week 6.
  The Modified Oswestry Disability Index, a condition specific questionnaire covering 10 areas of daily living and expressing the degree of disability as a percentage. The measured areas include: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment. Each category is scored on a continuum from 0 to 5 points, for a possible total score of 50 out of 50, popularly described as "100% disability."

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | This outcome will also be collected at secondary time points which include additional bi-weekly time points during care at Weeks 2, 4, 8, 10, and 12; as well as, 3, 6, and 12 months post-care.
Modified Oswestry Disability Index (MODI) | This outcome will also be collected at secondary time points which include additional bi-weekly time points during care at Weeks 2, 4, 8, 10, and 12; as well as, 3, 6, and 12 months post-care.

CONTACTS AND LOCATIONS:
Overall Officials: Jerrilyn Cambron, DC, MPH, PhD, Principal Investigator — National University of Health Sciences
Locations (1):
- National University of Health Sciences, Lombard, Illinois, United States

REFERENCES:
- [Derived] Cambron JA, Dexheimer JM, Duarte M, Freels S. Shoe Orthotics for the Treatment of Chronic Low Back Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Sep;98(9):1752-1762. doi: 10.1016/j.apmr.2017.03.028. Epub 2017 Apr 30. PMID 28465224